CLINICAL TRIAL: NCT04590924
Title: Pain, Function and Hip Osteoarthritis 5 Years After Hip Arthroscopic Surgery in Patients With Femoroacetabular Impingement
Brief Title: HAFAI Cohort 5 Year Follow up of Patients With Femoroacetabular Impingement Undergoing Hip Arthroscopy
Status: Completed | Type: Observational
Sponsor: Horsens Hospital (Other)
Responsible Party: Principal Investigator, Jeppe Lange, Primary investigator, Horsens Hospital
Other Study IDs: 1-10-72-1-19
Record Dates: First submitted 2019-09-04; First posted 2020-10-19 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Femoro Acetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hip arthroscopy — Patients that had hip arthroscopic surgery 5 years ago will be invited for 5 year follow up. The surgical procedures consisted of femoral osteoplasty, labral refixation and acetabular osteoplasty

SUMMARY:
Patients included in the HAFAI cohort will be invited for 5 year follow up.

DETAILED DESCRIPTION:
Patients with femoroacetabular impingement will be investigated 5 years after surgery. We will used the Copenhagen Hip and Groin Score to evaluate pain, activities of daily living, sport, participation in sport and hip-related quality of life. Furthermore, degree of hip osteoarthritis will be evaluated using standing x-rays. Last, we will investigate number of re-operations and conversions to total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Included in the HAFAI cohort

Exclusion Criteria:

* Non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the HAFAI cohort 5 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Pain 5 years after surgery | Score at 5 years and change from before surgery to 5 years after surgery
  Pain 5 years after surgery measured with the Copenhagen hip and groin scale (0-100 score)
Sports function 5 years after surgery | Score at 5 years and change from before surgery to 5 years after surgery
  Sports function 5 years after surgery measured with the Copenhagen hip and groin scale (0-100 score)
Development of osteoarthritis 5 years after surgery | Score at 5 years and change from before surgery to 5 years after surgery
  Lateral hip joint space width measured at anterior posterior standing radiographs
Re-operation | From date of initial surgery until the date of first documented re-operation or total hip replacement, whichever came first, assessed up to 6 years after initial surgery
  Re-operation/total hip replacement

SECONDARY OUTCOMES:
Activities of daily living 5 years after surgery | Score at 5 years and change from before surgery to 5 years after surgery
  Activities of daily living 5 years after surgery measured with the Copenhagen hip and groin scale (0-100 score)
Hip related quality of life 5 years after surgery | Score at 5 years and change from before surgery to 5 years after surgery
  Hip related quality of life 5 years after surgery measured with the Copenhagen hip and groin scale (0-100 score)
Participation in sport 5 years after surgery (HAGOS) | Score at 5 years and change from before surgery to 5 years after surgery
  Participation in sport 5 years after surgery measured with the Copenhagen hip and groin scale (0-100 score)
Participation in sport 5 years after surgery (HSAS) | Score at 5 years and change from before surgery to 5 years after surgery
  Participation in sport 5 years after surgery measured with Hip Sports activity scale

CONTACTS AND LOCATIONS:
Overall Officials: Signe Kierkegaard, PhD, Principal Investigator — Horsens Hospital
Locations (1):
- Signe Kierkegaard, Horsens, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kierkegaard S, Mechlenburg I, Dalgas U, Lund B. Five-Year Follow-up After Hip Arthroscopic Surgery in the Horsens-Aarhus Femoroacetabular Impingement (HAFAI) Cohort. Orthop J Sports Med. 2022 Mar 8;10(3):23259671221075653. doi: 10.1177/23259671221075653. eCollection 2022 Mar. PMID 35284589